CLINICAL TRIAL: NCT01261897
Title: The Efficacy of Adductor-Canal-Blockade on Pain and Morphine Consumption After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pia Jaeger, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM2-PJ-10; 2010-021918-30 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Postoperative Pain; Knee Arthroplasty
Keywords: Adductor-Canal-Blockade; postoperative pain; US-guided nerve block; total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adductor-Canal-Blockade with Ropivacaine (Active Comparator)
  Interventions: Procedure: Adductor-Canal-Blockade with Ropivacaine
- Adductor-Canal-blockade with saline (Placebo Comparator)
  Interventions: Procedure: Adductor-Canal-blockade with saline

INTERVENTIONS:
Procedure: Adductor-Canal-Blockade with Ropivacaine — US-guided Adductor-Canal-Blockade with ropivacaine 7,5 mg/ml
  Other Names: Naropine; Postoperative pain; US-guided nerve block
  Arms: Adductor-Canal-Blockade with Ropivacaine
Procedure: Adductor-Canal-blockade with saline — US-guided Adductor-Canal-blockade with saline
  Other Names: Sham block
  Arms: Adductor-Canal-blockade with saline

SUMMARY:
The objective of this study is to assess the efficacy of Adductor-Canal-Blockade on pain and morphine consumption after total knee arthroplasty. Our hypothesis is that the Adductor -Canal-Blockade is superior to placebo in reducing pain and morphine consumption after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Total Knee Arthroplasty in general anaesthesia
* ASA 1-3
* BMI 18-40
* Written informed consent

Exclusion Criteria:

* Can not cooperate to the exam
* Do not speak or understand Danish
* Drug allergy
* Alcohol or drug abuse
* Daily consumption of strong opioids

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pain during 45 degrees active flexion of the knee | 1 hour postoperative
  0-100 mm at a visual analogue scale (VAS), at 1 hour postoperative

SECONDARY OUTCOMES:
Pain during 45 degrees active flexion of the knee | 0-6 hours postoperative
  0-100 mm at a visual analogue scale (VAS), registered at the intervals 1, 2, 3, 4, 5 and 6 hours postoperative, calculated as "the area under the curve" (AUC) for the interval 1-6 hours postoperative.
Pain during rest | 1-6 hours postoperative
  0-100 mm at a visual analogue scale (VAS), registered at the intervals 1, 2, 3, 4, 5 and 6 hours postoperative, calculated as "the area under the curve" (AUC) for the interval 1-6 hours postoperative.
A change in pain score in the ropivacaine group, after activating the block | 30-60 minutes postoperative
  0-100 mm at a visual analogue scale (VAS), at 30 and 60 minutes postoperative. A change in pain score in the ropivacaine group compared to the placebo group, after activating the block.
Total morphine consumption | 30 minutes - 6 hours postoperative
  Total morphine consumption at the interval 30 minutes - 6 hours postoperative.
Postoperative nausea | 1-6 hours postoperative
  Nausea scores(0-3)registered at 1, 2, 3, 4, 5 and 6 hours postoperative, calculated as mean value for the interval 1-6 hours postoperative.
Postoperative vomiting | 1-6 hours postoperative
  Number of vomiting episodes at the interval 1-6 hours postoperative.
Zofran consumption | 1-6 hours postoperative
  Total zofran consumption at the intervals 1-6 hours postoperative.
Sedation | 1-6 hours postoperative
  Sedation score (0-3) registered at 1, 2, 3, 4, 5 and 6 hours postoperative, calculated as the mean value for the interval 1-6 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jæger, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Anaesthesia-Surgery-Intensive Care, Gentofte Hospital, Gentofte Municipality, Hellerup, Denmark

REFERENCES:
- [Derived] Jaeger P, Grevstad U, Henningsen MH, Gottschau B, Mathiesen O, Dahl JB. Effect of adductor-canal-blockade on established, severe post-operative pain after total knee arthroplasty: a randomised study. Acta Anaesthesiol Scand. 2012 Sep;56(8):1013-9. doi: 10.1111/j.1399-6576.2012.02737.x. Epub 2012 Jul 26. PMID 22834681